CLINICAL TRIAL: NCT01137656
Title: Storage Lesion in Banked Blood Due to Disruption of Nitric Oxide (NO) Homeostasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mark Gladwin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Mark Gladwin, Division Chief, Pulmonary, Allergy and Critical Care Medicine University of Pittsburgh Medical Center / Director, Vascular Medicine Institute of the University of Pittsburgh, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 686; R01HL098032-01 (NIH)
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: Blood storage; Blood transfusion; Aged blood; Blood Forearm; Storage lesion in blood
MeSH Terms: interventions — Acetylcholine; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acetylcholine and Blood (Other): This is single arm study. Acetylcholine and blood is infused in brachial artery of non-dominant arm. Blood flow
  Interventions: Drug: Acetylcholine and Blood

INTERVENTIONS:
Drug: Acetylcholine and Blood — The Acetylcholine solution will be infused intra-arterially at the dosage of 7.5 ug/min for 3 minutes, then 15ug/min for 3 minutes, then 30 ug/min for 3 minutes, after the infusion of normal saline. It will then be infused at 7.5ug/min for 3 minutes, followed by 15ug/min for 3 minutes, followed by 30 ug/min for 3 minutes after the infusion of autologous blood. This will be performed at 5-10 days and 35-42 days of blood storage time.
  Other Names: Miochol-e; Miochol

SUMMARY:
The purpose of this study is to explore the impact of aged blood on endothelial function by measuring forearm blood flow during intra-arterial acetylcholine infusion in normal healthy human volunteers after infusion of autologous blood stored for 5-10 days or 35-42 days.

Our hypothesis is that 1) the vasodilatory response to the infusion of acetylcholine will be reduced in the 35-42 day group compared with the 5-10 day group, because of scavenging of the NO released from the endothelium by the hemolytic process in the aged blood, 2) that the infusion of aged stored blood will produce vasoconstriction, measured by reduced forearm blood flow during infusion of the 35-42 day compared with the 5-10 day old blood, and that 3) there will be increases in venous levels of cell free plasma hemoglobin, red cell microparticles, red cell membrane damage, arginase levels and activity, decreased arginine levels, markers of oxidative stress (carbamylated proteins and nitrated tyrosine residues), and increases in plasma in vitro NO consumption during the infusion of 35-42 day old compared to 5-10 day old blood.

DETAILED DESCRIPTION:
The increased storage time of transfused blood is associated with an increased risk of cardiovascular events and organ failure. The underlying biological mechanism as to why this happens is not understood. A major abnormality in aged blood is the reduced life span of red blood cells after they are infused. This is associated with rupture of the red blood cells and release of their contents. However, the degree of red blood cell rupture and release of the cell's contents in humans after transfusion has not been well studied. It has been seen that even low levels of red blood cell rupture severely decrease the amount of nitric oxide and other factors that effect how blood vessels function. The purpose of this study is to perform human forearm blood flow studies to evaluate wether there are a sufficient amount these factors released during red blood transfusion to significantly affect how blood vessel function in humans.

This study will enroll normal healthy volunteers between 18 to 50 years of age. 500 ml (1.0 unit) of blood will be collected from subjects who will then return in 5-10 days and be re-infused with the blood 5-10 days after storage.The subjects will return after 25-37 days and be infused with blood 35-42 days after storage. The study will use a tool called strain gauge plethysmography and the drug acetylcholine to measure the effect of fresh (i.e., 5-10 days) versus aged (35-42 days) autologous blood transfusions on forearm blood flow in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and 18 to 50 years of age.
* Able to read and comprehend the English language

Exclusion Criteria:

* Less than 18 or greater than 50 years of age.
* Female < 110 lbs or 50 kg
* Male < 110 lbs or 50 kg
* Hemoglobin <12.5g/dl
* Past medical history or symptoms of blood dyscrasia, diabetes mellitus, hyperlipidemia, obstructive sleep apnea, hypertension, significant cardiac disease and / or known peripheral arterial disease.
* History of cigarette smoking within the last month
* Serum creatinine >1.0 mg/dL
* Cognitively impaired subjects, or institutionalized persons and subjects unable or unwilling to complete written informed consent (no proxy consent will be obtained)
* Subjects with a history of blood donation within the last 60 days.
* Subjects who have performed other medical studies involving drug delivery in the last 30 days.
* Subjects with an oxygen saturation value < 92%.
* Any STATIN drug (Fluvastatin, Lovastatin, Pravastatin, Simvastatin, Rosuvastatin) currently or in the 4 weeks prior to the screening day
* Any medication for the treatment of diabetes including oral hypoglycemics or insulin
* lab tests indicating blood dyscrasia, diabetes, hypertension or hypercholesterolemia.Females of childbearing potential who are pregnant or unwilling to undergo pregnancy testing; females with positive pregnancy testing on screening day will be excluded

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2010-04; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Blood flow response to Acetylcholine. | 5-10 days vs 35-42 days
  The primary endpoint will be a comparison of the blood flow responses to the acetylcholine after infusion of 5-10 day old blood compared with the responses after infusion of 35-42 day old blood, each controlled for the opposite arm.

SECONDARY OUTCOMES:
Change in blood flow response to fresh blood (5-10 days) in comparison to aged blood. | 5-10 days vs 35-42 days
  A comparison of the change in blood flow responses at baseline and after infusion of 5-10 day old blood compared with the responses during infusion of 35-42 day old blood, each controlled for the opposite arm.
Comparison in the levels of various biomarkers of aged blood will be examined in venous blood collected from the antecubital vein during the infusion of 5-10 days versus35-42 days old autologous blood. | 5-10 days versus 35-42 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Gladwin, M.D, Principal Investigator — University of Pittsburgh and University of Pittsburgh medical center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Greenwalt TJ, Bryan DJ, Dumaswala UJ. Erythrocyte membrane vesiculation and changes in membrane composition during storage in citrate-phosphate-dextrose-adenine-1. Vox Sang. 1984;47(4):261-70. doi: 10.1111/j.1423-0410.1984.tb01596.x. PMID 6485302
- [Background] Rumsby MG, Trotter J, Allan D, Michell RH. Recovery of membrane micro-vesicles from human erythrocytes stored for transfusion: a mechanism for the erythrocyte discocyte-to-spherocyte shape transformation. Biochem Soc Trans. 1977;5(1):126-8. doi: 10.1042/bst0050126. No abstract available. PMID 892138
- [Background] Dern RJ, Brewer GJ, Wiorkowski JJ. Studies on the preservation of human blood. II. The relationship of erythrocyte adenosine triphosphate levels and other in vitro measures to red cell storageability. J Lab Clin Med. 1967 Jun;69(6):968-78. No abstract available. PMID 6025497
- [Background] Berezina TL, Zaets SB, Morgan C, Spillert CR, Kamiyama M, Spolarics Z, Deitch EA, Machiedo GW. Influence of storage on red blood cell rheological properties. J Surg Res. 2002 Jan;102(1):6-12. doi: 10.1006/jsre.2001.6306. PMID 11792145
- [Derived] Risbano MG, Kanias T, Triulzi D, Donadee C, Barge S, Badlam J, Jain S, Belanger AM, Kim-Shapiro DB, Gladwin MT. Effects of Aged Stored Autologous Red Blood Cells on Human Endothelial Function. Am J Respir Crit Care Med. 2015 Nov 15;192(10):1223-33. doi: 10.1164/rccm.201501-0145OC. PMID 26222884